CLINICAL TRIAL: NCT03763318
Title: A Phase 1b/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of EQ001 in Subjects With Newly Diagnosed Acute Graft Versus Host Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, PK, PD, and Clinical Activity of EQ001 in Subjects With aGVHD
Acronym: EQUATE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Equillium (Industry)
Collaborators: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EQ001-aGVHD-001
Record Dates: First submitted 2018-11-19; First posted 2018-12-04 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Acute-graft-versus-host Disease; aGVHD; GVHD; GVHD, Acute
MeSH Terms: conditions — Graft vs Host Disease | interventions — itolizumab

STUDY DESIGN:
Intervention Model Description: Part A is an open label 3+3 dose escalation Part B is blinded and randomized 2:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part B will be blinded to all study staff that has direct access to the subjects and the sponsor. The site's pharmacist or designee will be unblinded to prepare the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EQ001 Dose Escalation (Part A) (Experimental): Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses.
  Interventions: Biological: EQ001
- EQ001 (Part B) (Experimental): EQ001 administered in a blinded fashion using the optimal dose selected from Part A by intravenous infusion every two weeks for a total of 5 doses.
  Interventions: Biological: EQ001
- EQ001 Placebo (Part B) (Placebo Comparator): Placebo administered in a blinded fashion by intravenous infusion every two weeks for a total of 5 doses.
  Interventions: Biological: EQ001 Placebo

INTERVENTIONS:
Biological: EQ001 — Itolizumab [Bmab 600])
  Other Names: Bmab600; Itolizumab
  Arms: EQ001 (Part B); EQ001 Dose Escalation (Part A)
Biological: EQ001 Placebo — EQ001 Placebo
  Arms: EQ001 Placebo (Part B)

SUMMARY:
This is a multi-center study to evaluate the safety, tolerability, PK, PD, and clinical activity of EQ001 in subjects with Acute Graft Versus Host Disease (aGVHD).

DETAILED DESCRIPTION:
The study will enroll approximately 100 subjects in two (2) parts:

Part A is an open label study and will enroll approximately 40 evaluable subjects with aGVHD across 4 cohorts. The total number of patients will depend on the number of dose escalations necessary to enable a decision to be made on the recommended dose to take forward into Part B of the study. The planned dose escalation will start with cohort 1, where subjects will receive EQ001 administered intravenously every two weeks for a total of 5 doses.

Part B is a randomized, double-blind, placebo-controlled study and will enroll approximately 60 additional subjects, randomized in a 2:1 ratio to either active treatment EQ001 (40) or placebo (20). Subjects will receive either EQ001 or placebo administered intravenously every two weeks for a total of 5 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject at least 18 years of age for Part A, and at least 12 years of age for Part B.
2. Recipients of allogeneic hematopoietic stem cell transplantation (alloHSCT) using myeloablative or non myeloablative conditioning regimens.
3. Have a clinical diagnosis of acute GVHD requiring systemic immune suppressive therapy.
4. Deemed by the investigator to be likely to comply with the planned procedure as required by the protocol for the duration of the study

Exclusion Criteria:

1. Presence of morphologic relapsed primary malignancy, treatment for relapse after alloHSCT was performed, or requirement for rapid immunosuppressive treatment withdrawal for early malignancy relapse.
2. Evidence of graft failure based on cytopenia(s), and as determined by the investigator.
3. Evidence of post-transplant lymphoproliferative disease.
4. Any prior therapy for acute GVHD, except for alloHSCT prophylaxis regimens or systemically administered corticosteroids.
5. As determined by the investigator, any medical, psychiatric, or other condition or circumstance that is likely to negatively affect: the subject's participation in this clinical study, the subject's safety, or the reliability of the study data.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Rothman, Study Director — Equillium
Locations (16):
- United States (16):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University and Barnes Jewish Heart & Vascular Center, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - TriStar Centennial Medical Center (SCRI), Nashville, Tennessee
  - Intermountain Healthcare, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rambaldi B, Kim HT, Arihara Y, Asano T, Reynolds C, Manter M, Halpern M, Weber A, Koreth J, Cutler C, Gooptu M, Nikiforow S, Ho VT, Antin JH, Romee R, Ampudia J, Ng C, Connelly S, Soiffer RJ, Ritz J. Phenotypic and functional characterization of the CD6-ALCAM T-cell co-stimulatory pathway after allogeneic cell transplantation. Haematologica. 2022 Nov 1;107(11):2617-2629. doi: 10.3324/haematol.2021.280444. PMID 35484649
- See also: Company website — https://equilliumbio.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part B of the study was not conducted.
Groups:
- EQ001 Dose Escalation (Part A) 0.4mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.4mg/kg
  EQ001: Itolizumab [Bmab 600]
- EQ001 Dose Escalation (Part A) 0.8mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.8mg/kg
  EQ001: Itolizumab [Bmab 600]
- EQ001 Dose Escalation (Part A) 1.6mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 1.6mg/kg
  EQ001: Itolizumab [Bmab 600]
Period: Overall Study
Arm/Group | EQ001 Dose Escalation (Part A) 0.4mg/kg | EQ001 Dose Escalation (Part A) 0.8mg/kg | EQ001 Dose Escalation (Part A) 1.6mg/kg
Started | 4 | 17 | 9
Completed | 3 | 7 | 3
Not Completed | 1 | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EQ001 Dose Escalation (Part A) 0.4mg/kg | EQ001 Dose Escalation (Part A) 0.8mg/kg | EQ001 Dose Escalation (Part A) 1.6mg/kg | Total
Number analyzed (Participants) | 4 | 17 | 9 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (18.03) | 60.1 (10.86) | 54.6 (12.98) | 56.3 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 4 | 10
  Male | 4 | 11 | 5 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 3
  White | 4 | 14 | 8 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of participants with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time Frame: Study Day 85
Measure: Count of Participants; unit: Participants
Groups:
- EQ001 Dose Escalation (Part A) 0.4mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.4mg/kg
  EQ001: Itolizumab [Bmab 600])
- EQ001 Dose Escalation (Part A) 0.8mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.8mg/kg
  EQ001: Itolizumab [Bmab 600])
- EQ001 Dose Escalation (Part A) 1.6mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 1.6mg/kg
  EQ001: Itolizumab [Bmab 600])
Arm/Group | EQ001 Dose Escalation (Part A) 0.4mg/kg | EQ001 Dose Escalation (Part A) 0.8mg/kg | EQ001 Dose Escalation (Part A) 1.6mg/kg
Number analyzed (Participants) | 4 | 17 | 9
Participants | 4 | 17 | 9

2. Primary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) is defined as the number of subjects with a partial response (PR), very good partial response (VGPR), or complete response (CR) who are alive at Day 29. Subjects must not have received new systemic therapy for aGVHD before the Day 29 Visit.
Time Frame: Study Day 29
Measure: Count of Participants; unit: Participants
Groups:
- EQ001 Dose Escalation (Part A) 0.4mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.4mg/kg.
  EQ001: Itolizumab [Bmab 600])
- EQ001 Dose Escalation (Part A) 0.8mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.8mg/kg.
  EQ001: Itolizumab [Bmab 600])
- EQ001 Dose Escalation (Part A) 1.6mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 1.6mg/kg.
  EQ001: Itolizumab [Bmab 600])
Arm/Group | EQ001 Dose Escalation (Part A) 0.4mg/kg | EQ001 Dose Escalation (Part A) 0.8mg/kg | EQ001 Dose Escalation (Part A) 1.6mg/kg
Number analyzed (Participants) | 4 | 17 | 9
Participants | 2 | 10 | 5

3. Secondary Outcome: Time to Maximum EQ001serum Concentration, Tmax
Description: Time to maximum EQ001 serum concentration, Tmax
Time Frame: Day 337
Reporting Status: Not Posted

4. Secondary Outcome: Maximum EQ001 Serum Drug Concentration, Cmax
Description: Maximum EQ001 serum drug concentration, Cmax
Time Frame: Study Day 337
Reporting Status: Not Posted

5. Secondary Outcome: Minimum EQ001 Serum Drug Concentration, Cmin
Description: Minimum EQ001 serum drug concentration prior to next dose, Cmin
Time Frame: Study Day 337
Reporting Status: Not Posted

6. Secondary Outcome: Total EQ001 Exposure Across Time, AUC (From Zero to Infinity)
Description: Total EQ001 exposure across time, AUC (from zero to infinity)
Time Frame: Study Day 337
Reporting Status: Not Posted

7. Secondary Outcome: Half Life of EQ001, t1/2
Description: Half life of EQ001, t1/2
Time Frame: Study Day 337
Reporting Status: Not Posted

8. Secondary Outcome: Volume of Distribution of EQ001, Vd
Description: Volume of distribution of EQ001, Vd
Time Frame: Study Day 337
Reporting Status: Not Posted

9. Secondary Outcome: Clearance, Cl
Description: Clearance, Cl
Time Frame: Study Day 337
Reporting Status: Not Posted

10. Secondary Outcome: Inflammatory Markers
Description: Including but not limited to: IL-1β, IL-2, IL-6, IL-17, IL-21, IL-22, IL-23, IFN-γ, and TGF-β, C-reactive protein
Time Frame: Study Day 337
Reporting Status: Not Posted

11. Secondary Outcome: CD6 Receptor Expression Levels
Description: CD6 receptor expression levels - percent of baseline
Time Frame: Study Day 85
Measure: Mean (Standard Deviation); unit: Percent of baseline
Groups:
- EQ001 Dose Escalation (Part A) 0.4mg/kg: Open label EQ001 administered by intravenous infusion every 14 days for a total of 5 doses at 0.4mg/kg.
  EQ001: Itolizumab [Bmab 600])
- EQ001 Dose Escalation (Part A) 0.8mg/kg: Open label EQ001 administered by intravenous infusion every 14 days for a total of 5 doses at 0.8mg/kg.
  E001: Itolizumab [Mab 600]
- Eq001 Dose Escalation (Part A) 1.6mg/kg: Open label EQ001 administered by intravenous infusion every 14 days for a total of 5 doses at 1.6mg/kg.
  E001: Itolizumab [Mab 600]
Arm/Group | EQ001 Dose Escalation (Part A) 0.4mg/kg | EQ001 Dose Escalation (Part A) 0.8mg/kg | Eq001 Dose Escalation (Part A) 1.6mg/kg
Number analyzed (Participants) | 4 | 17 | 9
Percent of baseline | 81.0 (17.78) | 23.7 (15.76) | 33.0 (19.25)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signing of the informed consent form through the long-term follow-up visit at Day 337.
Groups:
- EQ001 Dose Escalation (Part A) 0.4mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.4mg/kg.
  EQ001: Itolizumab [Bmab 600]
- EQ001 Dose Escalation (Part A) 0.8mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 0.8mg/kg.
  EQ001: Itolizumab [Bmab 600]
- EQ001 Dose Escalation (Part A) 1.6mg/kg: Open label EQ001 administered by intravenous infusion every two weeks for a total of 5 doses at 1.6mg/kg.
  EQ001: Itolizumab [Bmab 600]
Arm/Group | EQ001 Dose Escalation (Part A) 0.4mg/kg | EQ001 Dose Escalation (Part A) 0.8mg/kg | EQ001 Dose Escalation (Part A) 1.6mg/kg
All-Cause Mortality (participants affected / at risk) | 1/4 | 7/17 | 6/9
Serious Adverse Events (participants affected / at risk) | 2/4 | 9/17 | 8/9
Other Adverse Events (participants affected / at risk) | 4/4 | 17/17 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQ001 Dose Escalation (Part A) 0.4mg/kg (N=4) | EQ001 Dose Escalation (Part A) 0.8mg/kg (N=17) | EQ001 Dose Escalation (Part A) 1.6mg/kg (N=9)
Sepsis (Infections and infestations) | 0 (0) | 9 (9) | 2 (2)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 8 (8)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nocardiosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
pulmonary mucormycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease (Immune system disorders) | 0 (0) | 3 (3) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis fulminant (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EQ001 Dose Escalation (Part A) 0.4mg/kg (N=4) | EQ001 Dose Escalation (Part A) 0.8mg/kg (N=17) | EQ001 Dose Escalation (Part A) 1.6mg/kg (N=9)
Oedema peripheral (General disorders) | 2 (2) | 9 (9) | 6 (6)
Fatigue (General disorders) | 1 (1) | 6 (6) | 3 (3)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 9 (9) | 3 (3)
Blood alkaline phosphate increased (Investigations) | 0 (0) | 4 (4) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (4) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood lactic acid increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Graft versus host disease (Immune system disorders) | 0 (0) | 3 (3) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 (1) | 1 (1) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperferritinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Corona virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haptoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BK virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus infection reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nocardiosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mucormycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin weeping (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Intensive care unit delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis fulminant (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Azoospermia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03763318/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT03763318/SAP_001.pdf